CLINICAL TRIAL: NCT02867826
Title: The Use of Cap-assisted Forward Viewing Endoscopy for Examination of the Ampulla of Vater
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Denise Peixoto Guimarães, Principal Investigator, Barretos Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BarretosCH - 20161
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Ampulla of Vater Intestinal-Type Adenoma
Keywords: Endoscopy; Ampulla of Vater; Duodenoscopy
MeSH Terms: interventions — Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cap-assisted endoscopy (Experimental): forward-viewing endoscope with a Cap attached at the tip
  Interventions: Device: Cap

INTERVENTIONS:
Device: Cap — Cap-assisted endoscopy

SUMMARY:
The aim of this study is to compare the visualization rates of the ampulla of Vater using forward- viewing endoscopes with or without cap attached to the distal end in the same patient.

DETAILED DESCRIPTION:
The complete visualization of the ampulla of Vater for the detection of ampullary neoplastic lesions is technically challenging with a forward-viewing endoscope. There are limited data in the relevant literature regarding the effectiveness of the Cap assisted forward viewing endoscope for accurate evaluation of the ampulla de Vater. Therefore, the aim of this study is to compare the visualization rates of the ampulla of Vater using forward-viewing endoscopes with or without cap attached to the distal end in the same patient.

ELIGIBILITY:
Inclusion Criteria:

* Cap-assisted endoscopy
* Referral to endoscopic examination of ampulla of Vater

Exclusion Criteria:

* Patients with surgically modified anatomy.
* Obstruction of the upper gastrointestinal tract.
* Contra-indication for endoscopy.
* Absence of informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visualization rates of the ampulla of Vater | Up to 30 minutes during gastrointestinal endoscopy

SECONDARY OUTCOMES:
Rates of complications for both groups. | Up to 3 hours after upper endoscopy
Additional time required for Cap-assisted endoscopy | Up to 30 minutes during upper endoscopy
Need for additional sedation required for the Cap-assisted endoscopy. | Up to 30 minutes during upper endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Denise P Guimarães, MD, PhD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva LC, Arruda RM, Botelho PFR, Taveira LN, Giardina KM, de Oliveira MA, Dias J, Oliveira CZ, Fava G, Guimaraes DP. Cap-assisted endoscopy increases ampulla of Vater visualization in high-risk patients. BMC Gastroenterol. 2020 Jul 9;20(1):214. doi: 10.1186/s12876-020-01361-5. PMID 32646369